CLINICAL TRIAL: NCT07391579
Title: Daily Tadalafil 5 mg Combined With On-Demand Sildenafil 100 mg for Treatment of Erectile Dysfunction in PDE-5I Non Responder Patients: A Multicenter Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Daily Tadalafil 5 mg Combined With On-Demand Sildenafil 100 mg for Treatment of Erectile Dysfunction in PDE-5I Non Responder Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Cairo University (Other); Ain Shams University (Other); Aswan University (Other); Luxor university (Other); Assiut University (Other); Minia University (Other); Alexandria University (Other); Tanta University (Other); October 6 University (Other); Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP.25.09.1039
Record Dates: First submitted 2025-11-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Erectile Dysfunctions
Keywords: Erectile Dysfunction; ED; Sildenafil; Tadalafil; PDE5i Non-Responders; Combination Therapy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Daily tadalafil 5 mg and on-demand sildenafil 100 mg
  Interventions: Drug: Tadalafil 5 mg & Sildenafil 100mg
- Group B (Placebo Comparator): daily Placebo and on demand sildenafil 100 mg
  Interventions: Drug: Sildenafil 100mg & placebo

INTERVENTIONS:
Drug: Tadalafil 5 mg & Sildenafil 100mg — daily dosing of Tadalafil 5 mg combined with on demand Sildenafil 100mg
  Arms: Group A
Drug: Sildenafil 100mg & placebo — Daily Placebo combined with on demand Sildenafil 100mg
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to evaluate whether daily dosing with tadalafil 5 mg combined with on-demand sildenafil 100 mg can improve erectile function in men with erectile dysfunction (ED) who do not respond to PDE5 inhibitor alone.

The main questions it aims to answer are:

* Does the combination of daily tadalafil and on-demand sildenafil lead to a greater improvement in erectile function (measured by the IIEF-EF domain) compared with on-demand sildenafil alone?
* Is the combination therapy safe and well tolerated in this patient population?

Researchers will compare:

* Group A: Daily tadalafil 5 mg plus on-demand sildenafil 100 mg
* Group B: Daily placebo plus on-demand sildenafil 100 mg

to determine whether the combination regimen provides superior improvement in erectile function and patient satisfaction.

Participants will:

* Undergo baseline assessment including medical history, physical examination, and laboratory tests.
* Be randomly assigned to one of the two treatment groups.
* Take the assigned medications for 12 weeks.
* Complete follow-up evaluations at 4, 8, and 12 weeks, including:

International Index of Erectile Function (IIEF-15) questionnaire Erection Hardness Score (EHS) assessment Reporting of any adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Sexually active male.
* History of ED for ≥6 months.
* Erectile function domain of IIEF-15 score <17.
* Documented failure to respond to PDE-5I [definition of non-responder patients are patients with ED who don't respond to maximum dose of PDE-5I on ≥4 occasions in spite of accurate timing and good sexual stimulation].
* Stable sexual relationship ≥ 6 months.

Exclusion Criteria:

* Penile anatomical deformities or Peyronie's disease.
* Pelvic surgery or radiation.
* Active malignancy or severe systemic illness.
* Previous penile surgery of any kind, such as penile prosthesis, penile lengthening, penile cancer surgery, penile plication or grafting.
* Contraindication to PDE5i (High risk cardiac patients, patients on nitrates, hypotension).
* Using other treatments for ED e.g., Intra-cavernoasl prostaglandin injection therapy.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in International Index of Erectile Function-5 (IIEF-5) total score | from baseline to 12 weeks after starting treatment
  The IIEF-5 is a validated 5-item questionnaire assessing erectile function, with total scores ranging from 5 to 25; higher scores indicate better erectile function.

SECONDARY OUTCOMES:
Change in Erection Hardness Score (EHS), assessed using the validated 4-point Erection Hardness Scale | from baseline to 12 weeks after starting treatment
  The Erection Hardness Score (EHS) is a validated 4-point scale assessing penile rigidity, with higher scores indicating better erectile hardness.
Change in International Index of Erectile Function (IIEF-15) total score | from baseline to 12 weeks after treatment
  The International Index of Erectile Function (IIEF-15) is a validated 15-item questionnaire assessing erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction, with total scores ranging from 5 to 75; higher scores indicate better sexual function.
Incidence and severity of adverse events graded according to CTCAE version 5.0 | from baseline up to 12 weeks after treatment
  Adverse events will be recorded at each follow-up visit and classified by type, severity, and relationship to the intervention. Severity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Shokeir, professor of urology, Study Chair — Urology & Nephrology Center, Masnoura university, Egypt
Locations (11):
- Egypt (11):
  - Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahlia Governorate
  - Faculty of medicine, Alexandria University, Alexandria
  - Faculty of medicine, Aswan university, Aswān
  - Faculty of Medicine - Assiut University, Asyut
  - Cairo University, faculty of medicine, Cairo
  - Faculty of medicine, Ain Shams University, Cairo
  - Faculty of medicine, Azhar University, Cairo
  - Faculty of medicine, october 6 Univeristy, Cairo
  - Faculty of medicine, Luxor university, Luxor
  - faculty of medicine, Minya University, Minya
  - Faculty of medicine, Tanta University, Tanta

IPD SHARING:
Plan to Share IPD: Undecided